CLINICAL TRIAL: NCT01203605
Title: European Surgical Outcomes Study: A Multi-centre, International Seven Day Evaluation of Patient Care and Clinical Outcomes for Patients Undergoing Non-cardiac Surgery
Brief Title: European Surgical Outcomes Study
Acronym: EuSOS
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: European Society of Anaesthesiology (Other); European Society of Intensive Care Medicine (Other)
Responsible Party: Dr Rupert Pearse, Queen Mary's University of London
Other Study IDs: EuSOS 1.1
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2011-06

CONDITIONS: Non-cardiac Surgery
Keywords: Operative surgical procedures; mortality; adverse effects; Postoperative complications; Epidemiological Study
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-patient adult non-cardiac surgery: Consecutive patients admitted to participating centres undergoing elective and non-elective non-cardiac surgery commencing during the seven day study period with a planned overnight stay. All eligible patients undergoing surgery within the seven day study period will be recruited wherever possible.

SUMMARY:
The European Surgical Outcomes Study (EuSOS) is a multi-centre, international cohort study of peri-operative care and clinical outcomes for patients undergoing non-cardiac surgery.

Participating centres throughout Europe will contribute routine clinical data describing all eligible patients who undergo surgery from 4th April 2011 to 11th April 2011. Patients will then be followed until hospital discharge (or for a maximum of 60 days) for duration of hospital stay and hospital mortality. Routine clinical data will also be collected for those patients admitted to critical care at any stage after surgery but during the same hospital admission. Specific objectives are to describe clinical outcomes and standards of peri-operative care for patients undergoing non-cardiac surgery in Europe.

DETAILED DESCRIPTION:
Research questions

1. What is the in-hospital mortality rate for patients undergoing non-cardiac surgery in Europe?
2. What is the duration of hospital stay for patients undergoing non-cardiac surgery in Europe?
3. What is the current standard of peri-operative critical care provision for patients undergoing non-cardiac surgery in Europe?
4. What is the current standard of haemodynamic (cardiac output) monitoring for patients undergoing non-cardiac surgery in Europe?
5. Is there any evidence of differences in the standard of peri-operative care provision for patients undergoing non-cardiac surgery in different health-care systems within Europe?
6. Is there any evidence of differences in hospital stay and mortality for patients undergoing major non-cardiac surgery in different health-care systems within Europe?
7. What factors determine planned and unplanned admission to critical care after surgery?
8. Are the factors associated with critical care admission similar to those associated with post-operative death?

Methods

International cohort study of all adult patients undergoing in-patient non-cardiac surgery from 4th April 2011 to 11th April 2011.

Centres

The investigators aim to recruit as many European centres as possible but anticipate that a minimum of 150 hundred centres in ten or more nations will be required.

Ethics approval

National co-ordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place. This study is in effect a large scale clinical audit. The investigators expect that in most, if not every participating country, there will be no requirement for individual patient consent as all data will be anonymised and is already recorded as part of routine clinical care.

Data collection

Data will be collected describing all eligible patients undergoing surgery within the seven day cohort period. These patients will then be followed up until hospital discharge. Data will then be fully anonymised and transcribed by local investigators onto an internet based electronic CRF. A centre specific form will be completed once for each hospital to provide data including university/non-university hospital, number of operating rooms, number and level of critical care beds, etc.

Data set

An operating room data sheet will be completed once for each patient recruited to include data describing patient factors (age, gender, American Society of Anesthesiologists grade, major co-morbid disease, etc), surgical factors (procedure category, grade and urgency of surgery, grade of surgeon, surgical checklist, etc), anaesthetic factors (anaesthetic technique, haemodynamic monitoring, airway, grade of anaesthetist, etc), post-operative care (post-operative recovery ward stay, post-operative invasive or non-invasive ventilation or inotrope within first 24 hours). A critical care data sheet will be completed once for each patient admitted to critical care at any time after surgery, to include data describing whether admission was planned or unplanned, organ support, SAPS III score and SOFA score etc). Patients will be followed until death or hospital discharge for the following outcomes: duration of critical care stay, critical care mortality, duration of hospital stay and in-hospital mortality.

Sample size calculation

The investigators anticipate that approximately 20,000 patients will be required to provide a sample of up to 2,000 admissions to critical care after surgery. Assuming an overall mortality rate following surgery of 1%, a sample size of 20,000 patients will yield 200 deaths. This will allow the inclusion of at least fifteen variables in a logistic regression model for mortality. The rate of admission to critical care is likely to vary between nations but an overall rate of 10% will yield data describing up to 2000 admissions to critical care, whilst an overall rate of 5% will yield 1000 admissions. This to allow construction of a robust logistic regression model for this outcome. 20,000 patients will also provide >99% confidence for the overall mortality rate with 0.37% confidence width. If 200 deaths are observed in an overall sample of 20,000 patients, the 99% confidence interval for the proportion would be (0.008 - 0.012) with a confidence width of 0.37%. This dataset would also have sufficient generalisability to inform the practice of peri-operative care on an international basis.

Statistical analysis

The data to be collected are all collected as part of routine clinical care. Categorical variables will be described as proportions and will be compared using chi-square or Fisher's exact test. Continuous variable will be described as mean and standard deviation if normally distributed or median and inter-quartile range if not normally distributed. Comparisons of continuous variables will be performed using one-way ANOVA or Mann-Whitney test as appropriate. Univariate analysis will be performed to test factors associated with planned and unplanned admission to critical care and / or in-hospital death. A multiple logistic regression model will be used to identify independent risk factors. A stepwise approach will be used to enter new terms into the logistic regression model where p<0.05 was set as the limit for inclusion of new terms. A logistic regression model will be performed to assess independent association between prognostic factors and outcomes. Results of logistic regression will be reported as adjusted odds ratios (OR) with 95% confidence intervals. A single final analysis is planned at the end of the study.

Organisation

The study will be conducted by the EuSOS study group on behalf of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. Local co-ordinators will lead in the EuSOS study in individual institutions ensuring all relevant regulatory approvals are in place and adequate training of staff. They will supervise data collection, ensure timely data return and act as guarantor for the integrity and quality of data collected.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to participating centres undergoing elective and non-elective non-cardiac surgery commencing during the seven day cohort period with a planned overnight stay

Exclusion Criteria:

* patients undergoing planned day-case surgery
* cardiac surgery
* neurosurgery
* radiological procedures
* obstetric procedures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In-patient adult non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 46985 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mortality | In-hospital (maximum 60 days)
  Mortality prior to actual hospital discharge regardless of location censored at 60 days.

SECONDARY OUTCOMES:
Duration of hospital stay | Within single hospital admission
  Time in days from day of surgery to actual hospital discharge regardless of location
Planned admission to critical care | Within same hospital admission
  Post-operative admission to critical care which was planned and agreed prior to surgery
Unplanned admission to critical care | Within same hospital admission
  Unplanned post-operative admission to critical care at any stage in the same hospital admission
Duration of critical care stay | Within same hospital admission
  Time in days from admission to critical care to actual discharge from critical care or death
28 day mortality | 28 days
  Mortality up to 28 days after primary surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Pearse, MBBS FRCA MD, Study Chair — Queen Mary's University of London, UK; Andrew Rhodes, MBBS FRCA, Principal Investigator — St Georges Hospital, London UK; Rui Moreno, MD, Principal Investigator — Hospital de Santo António dos Capuchos, Lisboa, Portugal; Paolo Pelosi, MD, Principal Investigator — University of Insubria, Varese, Italy.; Claudia Spies, MD, Principal Investigator — Charite University, Berlin, Germany; Jean-Louis Vincent, MD PhD, Principal Investigator — Erasme Hospital, Free University of Brussels, Belgium.; Benoit Vallet, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Lille, France.; Philip Metnitz, MD, Principal Investigator — Medizinische Universität Wien, Austria.; Peter Bauer, PhD, Principal Investigator — Medizinische Universität Wien, Austria.; Andreas Hoeft, MD PhD, Principal Investigator — University Hospital Bonn, Germany
Locations (28):
- National co-ordinator, Ghent, Belgium
- National co-ordinator, Zagreb, Croatia
- National co-ordinator, Nicosia, Cyprus
- National co-ordinator, Brno, Czechia
- National co-ordinator, Odense, Denmark
- National co-ordinator, Tallinn, Estonia
- National co-ordinator, Helsinki, Finland
- National co-ordinator, Nîmes, France
- National co-ordinator, Berlin, Germany
- National co-ordinator, Athens, Greece
- National co-ordinator, Pécs, Hungary
- National co-ordinator, Reykjavik, Iceland
- National co-ordinator, Mullingar, Ireland
- National co-ordinator, Udine, Italy
- National co-ordinator, Riga, Latvia
- National co-ordinator, Vilnius, Lithuania
- National co-ordinator, Leeuwarden, Netherlands
- National co-ordinator, Bergen, Norway
- National co-ordinator, Poznan, Poland
- National co-ordinator, Lisbon, Portugal
- National co-ordinator, Iași, Romania
- National co-ordinator, Belgrade, Serbia
- National co-ordinator, Košice, Slovakia
- National co-ordinator, Ljubljana, Slovenia
- National co-ordinator, Valladolid, Spain
- National co-ordinator, Malmo, Sweden
- National co-ordinator, Geneva, Switzerland
- National co-ordinator, London, United Kingdom

REFERENCES:
- [Derived] Ahmad T, Beilstein CM, Aldecoa C, Moreno RP, Molnar Z, Novak-Jankovic V, Hofer CK, Sander M, Rhodes A, Pearse RM. Variation in haemodynamic monitoring for major surgery in European nations: secondary analysis of the EuSOS dataset. Perioper Med (Lond). 2015 Sep 23;4:8. doi: 10.1186/s13741-015-0018-8. eCollection 2015. PMID 26405521
- [Derived] van Zaane B, van Klei WA, Buhre WF, Bauer P, Boerma EC, Hoeft A, Metnitz P, Moreno RP, Pearse R, Pelosi P, Sander M, Vallet B, Pettila V, Vincent JL, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Nonelective surgery at night and in-hospital mortality: Prospective observational data from the European Surgical Outcomes Study. Eur J Anaesthesiol. 2015 Jul;32(7):477-85. doi: 10.1097/EJA.0000000000000256. PMID 26001104
- [Derived] Jammer I, Ahmad T, Aldecoa C, Koulenti D, Goranovic T, Grigoras I, Mazul-Sunko B, Matos R, Moreno R, Sigurdsson GH, Toft P, Walder B, Rhodes A, Pearse RM; European Surgical Outcomes Study (EuSOS) group. Point prevalence of surgical checklist use in Europe: relationship with hospital mortality. Br J Anaesth. 2015 May;114(5):801-7. doi: 10.1093/bja/aeu460. Epub 2015 Jan 13. PMID 25586728
- [Derived] Baron DM, Hochrieser H, Posch M, Metnitz B, Rhodes A, Moreno RP, Pearse RM, Metnitz P; European Surgical Outcomes Study (EuSOS) group for Trials Groups of European Society of Intensive Care Medicine; European Society of Anaesthesiology. Preoperative anaemia is associated with poor clinical outcome in non-cardiac surgery patients. Br J Anaesth. 2014 Sep;113(3):416-23. doi: 10.1093/bja/aeu098. Epub 2014 May 14. PMID 24829444